CLINICAL TRIAL: NCT03320382
Title: Multiple Breath Washout in Paediatric Chronic Airways Disease: Building a Clinimetrics Dataset
Brief Title: Multiple Breath Washout, a Clinimetric Dataset
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 17/NI/0046
Record Dates: First submitted 2017-05-17; First posted 2017-10-25 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Cystic Fibrosis; Primary Ciliary Dyskinesia; Bronchiectasis; Asthma; Bronchitis; Sleep Disorder
MeSH Terms: conditions — Cystic Fibrosis; Ciliary Motility Disorders; Bronchiectasis; Asthma; Bronchitis; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Multiple breath washout testing — Multiple breath washout testing will be completed on different devices over time
  Other Names: Exhlayzer D (Ecomedics); Modified Innocor (Innovision); Amis 2000 (Respiratory Mass Spectrometer) (Innovision); EasyOne Pro (New Diagnostic Design (NDD) Medical Technologies Inc

SUMMARY:
Monitoring patients with chronic, inflammatory airways disease particularly in the early stages is hampered by the relative insensitivity of current outcome measures to detect subtle changes. Multiple breath washout is a potential sensitive test that is a useful readout of disease at these early stages but it lacks standardisation and knowledge of variability with reference to standard lung function measures. This is a Cross sectional and longitudinal observation study. The hypothesis is that multiple breath washout-derived indices will provide a robust signal of gas mixing inhomogeneity, correlating with conventional measures of airway disease severity. Multiple breath washout performed on different devices will generate indices which correlate but differ in value.

DETAILED DESCRIPTION:
Lung Clearance Index (LCI) has been shown to be more sensitive and perhaps more applicable in early stages of lung disease when compared to currently utilised physiological outcome measures, and yet it is not approved by regulatory agencies as a recognised surrogate outcome measure. This may highlight some of the lack of understanding within MBW; what is the best equipment to use, what is the minimal value of change to show an improvement in LCI, what is LCI's correlation with clinical outcome measures and what does the progression of LCI tell us about lung disease. These questions will be addressed with a view to contributing a body of data to guide decisions around its utility in both interventional drug trials and for monitoring in a clinical setting.

The aim of this study is to assess the suitability of LCI as a clinical outcome measure for both clinical trials and clinical monitoring of patients with inflammatory respiratory disease across the disease spectrum. Different testing modalities will be compared as well as assess the repeatability and validity of LCI for its determination as an outcome measure. Long-term follow up will allow an assessment of the relationship between LCI and future outcomes such as rate of decline in lung function and frequency of exacerbations, both recognised as relevant by regulatory agencies.

ELIGIBILITY:
Inclusion criteria

* For patients with the following respiratory disease, diagnosis confirmed by:
* CF: diagnosed by standard criteria
* PCD: diagnosed by ciliary beat frequency measurement, ciliary beat pattern analysis or electron microscopy of ciliary ultrastructure, or genetics
* Non-CF bronchiectasis: CT diagnosis of bronchiectasis and not fulfilling diagnostic criteria for CF or PCD
* Asthma: as diagnosed by standard diagnostic criteria of British Thoracic Society/Scottish Intercollegiate Guideline Network (BTS/SIGN) guidelines.
* Persistent bacterial bronchitis defined as a wet cough present for >1 month, usually with bronchoscopic evidence of chronic infection, that resolves with appropriate antibiotic therapy
* Sleep Disordered Breathing.
* For healthy volunteers, these will be colleagues and staff contacts (including children) at a participating centre i.e. Royal Brompton Hospital, or will be siblings of patients.
* Written informed consent (assent from children of appropriate age) obtained.

Exclusion criteria

* Positive culture (within the last year of / receiving treatment for Mycobaterium tuberculosis or abscessus (due to cross-infection concerns).
* Pregnant or breastfeeding.
* Inability to understand or cooperate with the test(s).
* Inability to give informed consent, or withdrawal of informed consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged two and upwards with chronic airways disease including CF, PCD, Asthma and Bronchiectasis, Persistent bacterial bronchitis and sleep disordered breathing and obesity as well as aged matched healthy control patients will be approached to take part in the study.
  Healthy volunteers will only complete MBW and Spirometry for comparison with respiratory disease patients.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Lung Clearance Index | Each testing session may take up to 90 minutes but most likely it will be under an hour. The MBW test will be completed at each visit and the LCI and other MBW results are obtained from data analysis post completion.
  Multiple breath washout involves recording concentrations of a tracer gas whilst it is cleared from the lungs during normal tidal breathing. The tracer gas can either be an inert gas such as sulphur hexafluoride (SF6) that is washed out by room air, or resident Nitrogen (N2) that is cleared by 100% oxygen (O2). All tracer gases are traditionally cleared to 1/40th (or 2.5%) of their starting concentration. This procedure is performed in triplicate, each test will take around 5-10 minutes with wait time in-between.

SECONDARY OUTCOMES:
Spirometry | Spirometry will be completed at each visit (unless already taken at a clinical visit). Maximum 10 visits over 3 years
  Spirometry is an effort dependant test designed to assess lung volumes.Spirometry will be performed according to ERS guidelines on a spirometer such as the Easyone with a disposable mouthpiece and filter. Three good quality measurements will be made and the best recorded in absolute values. Spirometry will only be collected in subjects age 6 and upwards (or if performed adequately at clinic visits at a younger age) since it is difficult to perform and produce reliable spirometry results in this young age
Disease specific Quality of life questionnaire | The quality of life questionnaire will be completed at each visit and compared to the primary outcome at each visit. Maximum 10 visits over 3 years
  Quality of Life Questionnaires provide patient-reported outcomes and how subjects are feeling in relation to new treatments or generally with regard to their lung disease. For certain diseases such as cystic fibrosis, these outcome measures are emerging as clinical tools, so it will not be duplicated if it has already been performed. A questionnaire will be completed either on paper or a computer at each visit to compare physiological data with how a patient is feeling.
  Validated Revised Cystic Fibrosis Questionnaire (CFQR) for CF patients. For Asthma patients, Paediatric Asthma Quality of life Questionnaire, Paediatric Asthma Caregivers Quality of Life Questionnaire, Asthma Control Test Score, Childhood Asthma Control Test score, Test for Respiratory and Asthma Control in Kids.
  For Primary Cilary Dyskinesia the new validated PCD questionnaire. Healthy volunteers will not complete a questionnaire.
Review of clinically indicated tests | Post each visit review of clinically indicated tests will take place and compared to the primary outcome. Maximum 10 visits over 3 years
  For patients with respiratory disease, some results taken for clinically indicated reasons either on the same day or close to the research day may be reviewed from clinical notes or hospital electronic data capture systems as part of this research for comparisons. These may include blood sample results, sputum cultures and clinically assessment from the multidisciplinary team within clinic letters.

CONTACTS AND LOCATIONS:
Overall Officials: Jane C Davies, Professor, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No